CLINICAL TRIAL: NCT02845440
Title: Integrated Smoking Cessation Treatment for Smokers With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bay Cove Human Services (Other); Brigham and Women's Hospital (Other); University of Massachusetts, Amherst (Other); Vinfen (Industry)
Responsible Party: Principal Investigator, A. Eden Evins, Director, Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P001036
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-02

CONDITIONS: Cigarette Smoking; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Smoking Cessation
Keywords: Pragmatic Trial; Community Health Workers; Academic Detailing
MeSH Terms: conditions — Cigarette Smoking; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Smoking Cessation | interventions — Community Health Workers; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment as Usual (TAU) - Cohort 1 (Active Comparator): Usual care (TAU) for adults with SMI in Massachusetts consists of rehabilitation services publicly funded by the state and traditional fee for service outpatient medical and psychiatric care. Importantly, medical care is not programmatically integrated with the psychiatric rehabilitation services. Participants in this arm will receive no other study-related intervention.Cohort 1 (AD-eligible) comprised participants seen in primary care clinics serving ≥3 enrolled participants.
  Interventions: Other: Treatment as Usual (TAU)
- AD + CHW - Cohort 1 (Experimental): Academic detailing (AD) is a targeted continuing medical education (CME) strategy that adapts social marketing techniques, using mixed interactive and didactic formats in individual and group settings integrated into the practice setting to promote beneficial changes in medical care. The aim of AD is to help clinicians understand and adopt targeted evidence-based practices.
  Community Health Worker (CHW) will offer to support patients and prescribers to implement smoking cessation treatments that may be requested by patients and/or recommended by prescribers.
  Interventions: Other: Academic Detailing; Other: Community Health Worker
- AD - Cohort 1 (Experimental): Participant in this arm will have Academic Detailing offered to their primary care clinical staff as described above. Participants who are randomized to this condition will not be offered Community Health Worker support.
  Interventions: Other: Academic Detailing
- CHW - Cohort 2 (Experimental): Community Health Worker (CHW) will offer to support patients and prescribers to implement smoking cessation treatments that may be requested by patients and/or recommended by prescribers.
  Interventions: Other: Community Health Worker
- Treatment as Usual (TAU) - Cohort 2 (Active Comparator): Usual care (TAU) for adults with SMI in Massachusetts consists of rehabilitation services publicly funded by the state and traditional fee for service outpatient medical and psychiatric care. Importantly, medical care is not programmatically integrated with the psychiatric rehabilitation services. Participants in this arm will receive no other study-related intervention. Cohort 2 (AD-ineligible) comprised participants whose primary care clinic served ≤2 enrolled participants
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: Academic Detailing — Academic detailing (AD) is a targeted continuing medical education (CME) strategy that adapts social marketing techniques, using mixed interactive and didactic formats in individual and group settings integrated into the practice setting to promote beneficial changes in medical care. AD helps clinicians understand and adopt targeted evidence-based practices and is one of the few Continuing Medical Education (CME) interventions that has consistently demonstrated improved alignment of physician prescribing behavior with evidence-based practice.
  Arms: AD + CHW - Cohort 1; AD - Cohort 1
Other: Community Health Worker — Community Health Worker (CHW) The CHW will offer to support patients and prescribers in health promotion and preventive care in general and specifically to support communication between the primary care provider and patient regarding smoking status, smoking cessation, and to aid implementation of any smoking cessation treatments recommended by prescribers. CHWs will complete the standard CHW certificate training program in general preventive medicine, available through the Boston Public Health Commission. CHWs will then receive the additional specialized training.
  Arms: AD + CHW - Cohort 1; CHW - Cohort 2
Other: Treatment as Usual (TAU) — Usual care (TAU) for adults with SMI in Massachusetts consists of rehabilitation services publicly funded by the state and traditional fee for service outpatient medical and psychiatric care. Importantly, medical care is not programmatically integrated with the psychiatric rehabilitation services.
  Arms: Treatment as Usual (TAU) - Cohort 1; Treatment as Usual (TAU) - Cohort 2

SUMMARY:
The overall aim of this study is to test the effect of academic detailing (i.e. provider-level educational intervention focused on evidence-based smoking cessation treatment for those with psychiatric illness) and community health worker (CHW) support on the provision and utilization of standard of care smoking cessation treatment to those with serious mental illness (SMI) and smoking cessation rates for adults with SMI who smoke.

DETAILED DESCRIPTION:
In this study, the investigators aim to test whether a provider-level educational intervention in the form of targeted, practical, action-oriented education to primary care physicians and nurses on safety and effectiveness of and how to use evidence-based smoking cessation treatment for those with psychiatric illness, termed academic detailing (AD), and practical support offered to the primary care physician / primary care team and the smoker with SMI in the form of a community health worker (CHW) will improve recommendation and utilization of standard of care smoking cessation treatments to and by those with SMI and, if so, whether the intervention improves smoking cessation rates for adults with SMI who smoke.

To do so, the investigators will enroll approximately 1300 adult smokers with SMI who receive psychiatric rehabilitation services, Community Based Flexible Support (CBFS) or Assertive Community Treatment (ACT)), from the two largest providers of these services in the Boston area. Primary care clinics that serve 3 or more enrolled participants will be cluster randomized in a 2:1 ratio to either receive AD for their clinical staff or treatment as usual (TAU) in a cluster randomized design. Smokers with SMI in the study who receive primary care at the clinics assigned to the AD intervention to providers will be randomly assigned at the individual level in a 1:1 ratio to be offered CHW support in addition to their ongoing psychiatric rehabilitation (CBFS or ACT) services. This was the original design for the study and these participants comprise Cohort 1. The protocol was modified and approved by the sponsor in February 2018 to include a second cohort. Because 155 enrolled participants received primary care in 155 clinics that served only 1-2 participants, and it was beyond the scope of the trial to deliver AD to so many clinics, a second cohort was formed in which these 155 participants were randomly assigned at the individual level in a 1:1 ratio to CHW or TAU.

This study was also modified by receipt of a qualitative supplement award from the sponsor to conduct mixed methods research to identify and define barriers and facilitators to implementation of components of the integrated care intervention in primary care clinical settings using an interactive convergent mixed-methods design. The aim of this portion of the study is to better understand the factors that impact the integration of Integrated Care and evidence-based treatments for smoking cessation for those with SMI in primary care settings. Qualitative interviews will be conducted for enrolled participants, CHWs, primary care physician, and stakeholders.

ELIGIBILITY:
Inclusion:

* adult (18+ years)
* current smoker
* current diagnosis of SMI (e.g. schizophrenia, bipolar disorder, major depressive disorder, etc...)
* currently receiving psychiatric rehabilitation services through CBFS and ACT programs at Bay Cove Human Services and Vinfen Corporation

Exclusion:

* intellectual disability (IQ<70)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1165 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Addiction Medicine, Massachusetts General Hospital, Dept. of Psychiatry, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Evins AE, Cather C, Maravic MC, Reyering S, Pachas GN, Thorndike AN, Levy DE, Fung V, Fischer MA, Schnitzer K, Pratt S, Fetters MD, Deeb B, Potter K, Schoenfeld DA. A Pragmatic Cluster-Randomized Trial of Provider Education and Community Health Worker Support for Tobacco Cessation. Psychiatr Serv. 2023 Apr 1;74(4):365-373. doi: 10.1176/appi.ps.20220187. Epub 2022 Nov 9. PMID 36349498

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual (TAU) Cohort 1: Usual care (TAU) for adults with SMI in Massachusetts consists of rehabilitation services publicly funded by the state and traditional fee for service outpatient medical and psychiatric care. Importantly, medical care is not programmatically integrated with the psychiatric rehabilitation services. Participants in this arm will receive no other study-related intervention.Cohort 1 (AD-eligible) comprised participants seen in primary care clinics serving ≥3 enrolled participants
- AD + CHW - Cohort 1: Academic Detailing: (AD) is a targeted continuing medical education strategy that adapts social marketing techniques, using mixed interactive and didactic formats in individual and group settings integrated into the practice setting to promote beneficial changes in medical care. AD helps clinicians understand and adopt targeted evidence-based practices and is one of the few Continuing Medical Education (CME) interventions that has consistently demonstrated improved alignment of physician prescribing behavior with evidence-based practice. The aim of AD is to help clinicians understand and adopt targeted evidence-based practices.
  Community Health Worker: (CHW) The CHW will offer to support patients and prescribers in health promotion and preventive care in general and specifically to support communication between the primary care provider and patient regarding smoking status, smoking cessation, and to aid implementation of any smoking cessation treatments recommended by prescribers. CHWs will complete the standard CHW certificate training program in general preventive medicine, available through the Boston Public Health Commission. CHWs will then receive the additional specialized training.
- AD - Cohort 1: Participants who are randomized to this condition will not be offered additional Community Health Worker services; however, the participant's primary care clinic will receive Academic Detailing
  Academic Detailing: Academic detailing (AD) is a targeted continuing medical education (CME) strategy that adapts social marketing techniques, using mixed interactive and didactic formats in individual and group settings integrated into the practice setting to promote beneficial changes in medical care. AD helps clinicians understand and adopt targeted evidence-based practices and is one of the few Continuing Medical Education (CME) interventions that has consistently demonstrated improved alignment of physician prescribing behavior with evidence-based practice.
- CHW - Cohort 2: Community Health Worker: (CHW) The CHW will offer to support patients and prescribers in health promotion and preventive care in general and specifically to support communication between the primary care provider and patient regarding smoking status, smoking cessation, and to aid implementation of any smoking cessation treatments that may be requested by patients and/or recommended by prescribers. CHWs will complete the standard CHW certificate training program in general preventive medicine, available through the Boston Public Health Commission. CHWs will then receive the additional specialized training.
- Treatment as Usual (TAU) Cohort 2: Usual care (TAU) for adults with SMI in Massachusetts consists of rehabilitation services publicly funded by the state and traditional fee for service outpatient medical and psychiatric care. Importantly, medical care is not programmatically integrated with the psychiatric rehabilitation services. Participants in this arm will receive no other study-related intervention.Cohort 2 (AD-ineligible) comprised participants whose primary care clinic served ≤2 enrolled participants.
Period: Overall Study
Arm/Group | Treatment as Usual (TAU) Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) Cohort 2
Started | 333 | 336 | 341 | 78 | 77
Completed | 201 | 203 | 204 | 49 | 39
Not Completed | 132 | 133 | 137 | 29 | 38

BASELINE CHARACTERISTICS:
Population: After enrollment completion, protocol was amended because 155 of 1165 particips received care at 111 clinics that served ≤2 particips. Providing AD to so many clinics was beyond the project scope, so, prior to randomization, it was decided (with sponsor approval) to include the 155 partics in cohort 2 in a stratified randomization: Cohort 1 (AD-eligible) with partics whose clinics served ≥3 partics. Cohort 2 (AD-ineligible) with partics whose clinic served ≤2 partics randomized to CHW or TAU
Groups:
- Treatment as Usual (TAU) Cohort 2: Cohort 2 (AD-ineligible) comprised participants whose primary care clinic served ≤2 enrolled participants. Usual care (TAU) for adults with SMI in Massachusetts consists of rehabilitation services publicly funded by the state and traditional fee for service outpatient medical and psychiatric care. Importantly, medical care is not programmatically integrated with the psychiatric rehabilitation services. Participants in this arm will receive no other study-related intervention.
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual (TAU) Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) Cohort 2 | Total
Number analyzed (Participants) | 333 | 336 | 341 | 78 | 77 | 1165
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (13.2) | 47.4 (12.7) | 47.3 (12.9) | 44.7 (14.2) | 46 (14.4) | 47.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 103 | 105 | 32 | 29 | 368
  Male | 234 | 233 | 236 | 46 | 48 | 797
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 60 | 69 | 19 | 9 | 199
  Not Hispanic or Latino | 291 | 276 | 272 | 59 | 68 | 966
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 149 | 165 | 158 | 59 | 52 | 583
  Black | 132 | 126 | 136 | 13 | 15 | 422
  Asian | 18 | 10 | 10 | 2 | 1 | 41
  Other | 17 | 11 | 11 | 1 | 3 | 43
  Multi-race | 17 | 24 | 26 | 3 | 6 | 76
Participants living in supervised Housing (Y/N) [Count of Participants; unit: Participants]
  Yes | 144 | 146 | 158 | 15 | 17 | 480
  No | 189 | 190 | 183 | 63 | 60 | 685
SF-1 M(SD) [Mean (Standard Deviation); unit: units on a scale] — The singe item self-reported Short Form Survey (SF-1) is used to assess health-related quality of life. It includes the following question: "In general, would you say your health is: Excellent (1), Very good (2), Good (3), Fair (4) or Poor (5)." Higher scores indicate worse health-related quality of life. The SF-1 has been validated as a descriptor of individual health and wellbeing as well as community health status.
  units on a scale | 3.1 (1.1) | 3.1 (1.1) | 3.2 (1.1) | 3.1 (1.1) | 3.2 (1.1) | 3.1 (1.1)
Expired Carbon Monoxide M(SD) [Mean (Standard Deviation); unit: ppm (parts per million)] | 25 (25.7) | 22.7 (18.5) | 22.6 (17.2) | 23.1 (19.4) | 20.9 (14.8) | 23.2 (20.3)
HSI M(SD) [Mean (Standard Deviation); unit: units on a scale] — The Heaviness of Smoking Index (HSI) is a composite measure that consists of 2 questions: number of cigarettes per day (CPD) assessed by: "On average, how many cigarettes do you smoke each day?" to provide a report of daily consumption, and for the standard HSI, the codes are 0: 1-10 CPD; 1: 11-20 CPD; 2: 21-30 CPD; and 3: 31+ CPD; and time to first cigarette (TTFC),ascertained by "How soon after waking do you usually have your first smoke?" Standard HSI codes are 0: 61+ min; 1: 31-60 min; 2: 6-30 min; and 3: ≤5 min. When summed, they give a scale with a range of 0-6.
  units on a scale | 2.9 (1.6) | 2.7 (1.6) | 2.9 (1.7) | 2.9 (1.6) | 3 (1.6) | 2.9 (1.6)
Number of Tobacco Products per day M(SD) [Mean (Standard Deviation); unit: products per day] | 15.7 (10.6) | 14.9 (9.6) | 16 (11.4) | 15.8 (9.7) | 15.5 (10.5) | 15.5 (10.5)
Participants that use Cigarettes %(n) [Count of Participants; unit: Participants] — Number that participants who reported smoking cigarettes at baseline
  Participants | 281 | 272 | 289 | 72 | 61 | 975
Participants that use Little cigars %(n) [Count of Participants; unit: Participants] — Number that participants who reported smoking little cigars at baseline
  Participants | 105 | 114 | 114 | 15 | 22 | 370
Participants that use Hand rolled cigarettes %(n) [Count of Participants; unit: Participants] — Number that participants who reported smoking hand rolled cigarettes at baseline
  Participants | 26 | 27 | 21 | 5 | 6 | 85
Participants that use E-cigarettes %(n) [Count of Participants; unit: Participants] — Number that participants who reported smoking e-cigarettes at baseline
  Participants | 6 | 1 | 8 | 2 | 4 | 21
Participants that received a Physician recommendation to quit smoking %(n) [Count of Participants; unit: Participants] | 231 | 205 | 217 | 49 | 47 | 749
Participants that were prescribed a medication to aid cessation %(n) [Count of Participants; unit: Participants] | 130 | 94 | 108 | 22 | 24 | 378
Participants that used Varenicline %(n) [Count of Participants; unit: Participants] | 30 | 17 | 14 | 3 | 2 | 66
Participants that used Bupropion %(n) [Count of Participants; unit: Participants] | 6 | 1 | 5 | 2 | 1 | 15
Participants that used Nicotine Replacement Therapy (any form) %(n) [Count of Participants; unit: Participants] | 124 | 89 | 99 | 20 | 23 | 355
Cardiovascular/respiratory illness %(n) [Count of Participants; unit: Participants] | 206 | 175 | 180 | 42 | 45 | 648
Other smoking related illness %(n) [Count of Participants; unit: Participants] | 40 | 36 | 44 | 13 | 14 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Abstinent at the Intervention Year 2 Assessment in Cohort 1
Description: Three pairwise comparisons between usual care (TAU), AD+CHW, and AD for number of participants who are abstinent (defined as 7-day point prevalence tobacco abstinence confirmed with an expired CO of 5 ppm or less) at the intervention year 2 assessment. The investigators hypothesize that (1) those who receive AD+CHW will demonstrate higher rates of tobacco abstinence than those who receive TAU, (2) those who receive AD will demonstrate higher rates of tobacco abstinence than those who received TAU, and (3) those who receive AD+CHW will demonstrate higher rates of tobacco abstinence than those who received AD.
Time Frame: Assessment at end of year 2 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1
Number analyzed (Participants) | 264 | 259 | 264
Participants | 13 | 32 | 19
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1; Missing data at year 2 of intervention was imputed using MICE based on baseline characteristics and outcome values at year 1 of intervention. The statistical model was a mixed effects logistic regression with terms for TAU, AD, and AD+CHW (cohort 1) and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Superiority; p = 0.013, Regression, Logistic — A priori threshold for significance was p < 0.05; Odds Ratio (OR) = 2.40, 95% CI 2-sided [1.20 to 4.79]
Statistical Analysis 2: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD - Cohort 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.481, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.62 to 2.74]
Statistical Analysis 3: Comparison: AD + CHW - Cohort 1 vs AD - Cohort 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.036, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.04 to 3.24]

2. Secondary Outcome: Number of Participants Who Use of Any First Line, Evidence-based TUD Medication at the Intervention Year 1 or 2 Assessment in Cohort 1
Description: Two comparisons, usual care (TAU) versus AD+CHW and TAU versus AD, for use of any first line, evidence-based TUD medication during assessments for years 1 and 2 of the intervention. The investigators hypothesize that (1) those who receive AD+CHW will demonstrate higher rates of medication use than those who received TAU, and (2) those who receive AD will demonstrate higher rates of medication use than those who received TAU.
Time Frame: Any use over assessments for years 1 or 2 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1
Number analyzed (Participants) | 264 | 259 | 264
Participants
  Any TUD med | 112 | 121 | 83
  No TUD med | 152 | 138 | 181
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1; The statistical model was a mixed effects logistic regression with terms for TAU, AD, and AD+CHW (cohort 1) and a clinic-varying random intercept; Test type: Superiority; p = 0.174, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.88 to 2.06]
Statistical Analysis 2: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD - Cohort 1; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.092, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.45 to 1.06]

3. Secondary Outcome: Number of Participants Who Use Varenicline at the Intervention Year 1 or 2 Assessment in Cohort 1
Description: Two comparisons, usual care (TAU) versus AD+CHW and TAU versus AD, for use of varenicline during assessments for years 1 and 2 of the intervention. The investigators hypothesize that (1) those who receive AD+CHW will demonstrate higher rates of varenicline use than those who received TAU, and (2) those who receive AD will demonstrate higher rates of varenicline use than those who received TAU.
Time Frame: Any use over assessments for years 1 or 2 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1
Number analyzed (Participants) | 264 | 259 | 264
Participants
  Varenicline | 34 | 72 | 30
  No varenicline | 230 | 187 | 234
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.61 to 4.75]
Statistical Analysis 2: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD - Cohort 1; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.742, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.50 to 1.64]

4. Secondary Outcome: Effect of Use of Any TUD Medication on Number of Participants Who Are Abstinence at the Intervention Year 2 Assessment in Cohort 1
Description: Effect of use of any first line, evidence-based TUD medication during assessments for years 1 and 2 of the intervention on number of participants who are abstinent (defined as 7-day point prevalence tobacco abstinence confirmed with an expired CO of 5 ppm or less) at the intervention year 2 assessment. The investigators hypothesize that those who used any medication will exhibit higher rates of tobacco abstinence than those who did not use any medications. The indirect effect of AD+CHW and AD interventions on abstinence rates with any TUD medication use as a mediator will be also be assessed.
Time Frame: Assessment at end of year 2 of intervention
Measure: Count of Participants; unit: Participants
Groups:
- AD - Cohort 1: Participants who are randomized to this condition will only not be offered additional Community Health Worker services; however, the participant's primary care clinic will receive Academic Detailing as described above.
  Academic Detailing: Academic detailing (AD) is a targeted continuing medical education (CME) strategy that adapts social marketing techniques, using mixed interactive and didactic formats in individual and group settings integrated into the practice setting to promote beneficial changes in medical care. AD helps clinicians understand and adopt targeted evidence-based practices and is one of the few Continuing Medical Education (CME) interventions that has consistently demonstrated improved alignment of physician prescribing behavior with evidence-based practice.
Arm/Group | Treatment as Usual (TAU) - Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1
Number analyzed (Participants) | 264 | 259 | 264
Participants
  Any TUD med + abstinent | 5 | 24 | 7
  No TUD med + abstinent | 8 | 8 | 12
  Any TUD med + not abstinent | 107 | 97 | 76
  No TUD med + not abstinent | 144 | 130 | 169
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD + CHW - Cohort 1 vs AD - Cohort 1; Missing abstinence rates at year 2 of intervention were imputed using MICE based on baseline characteristics and abstinence rates at year 1 of intervention. The statistical model was a mixed effects logistic regression with terms for TAU, AD, and AD+CHW (cohort 1) as well as TUD medication use and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Superiority; p = 0.056, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.99 to 2.51]; A mediation analysis found that the estimated proportion of the effect of TUD medication use on abstinence rates attributable to the AD+CHW intervention was 2.8%

5. Secondary Outcome: Effect of Varenicline Use on Number of Participants Who Are Abstinence at the Intervention Year 2 Assessment in Cohort 1
Description: Effect of use of varenicline during assessments for years 1 and 2 of the intervention on number of participants who are abstinent (defined as 7-day point prevalence tobacco abstinence confirmed with an expired CO of 5 ppm or less) at the intervention year 2 assessment. The investigators hypothesize that those who used varenicline will exhibit higher rates of tobacco abstinence than those who did not use any varenicline. The indirect effect of AD+CHW and AD interventions on abstinence rates with any TUD medication use as a mediator will be also be assessed.
Time Frame: Assessment at end of year 2 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) - Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1
Number analyzed (Participants) | 264 | 259 | 264
Participants
  Varenicline + abstinent | 1 | 17 | 4
  No varenicline + abstinent | 12 | 15 | 15
  Varenicline + not abstinent | 33 | 55 | 26
  No varenicline + not abstinent | 218 | 172 | 219
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD + CHW - Cohort 1 vs AD - Cohort 1; Missing abstinence rates at year 2 of intervention were imputed using MICE based on baseline characteristics and abstinence rates at year 1 of intervention. The statistical model was a mixed effects logistic regression with terms for TAU, AD, and AD+CHW (cohort 1) as well as varenicline use and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Superiority; p = 0.012, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.16 to 3.33]; A mediation analysis found that the estimated proportion of the effect of varenicline use on abstinence rates attributable to the AD+CHW intervention was 13.9%

6. Secondary Outcome: Number of Participants Who Are Abstinent at the Intervention Year 2 Assessment in Cohorts 1 and 2
Description: Comparisons between (1) CHW (pooled over AD+CHW and CHW) and (2) AD (pooled over AD+CHW and AD) compared to usual care (TAU) on number of participants who are abstinent (defined as 7-day point prevalence tobacco abstinence confirmed with an expired CO of 5 ppm or less) at the intervention year 2 assessment. The investigators hypothesize that (1) those who receive CHW support will demonstrate higher rates of tobacco abstinence than those who receive TAU, and (2) those with AD exposure will demonstrate higher rates of tobacco abstinence than those who received TAU. To make use of all the data, hypotheses will be assessed in Cohorts 1 and 2 via analysis of a factorial design.
Time Frame: Assessment at end of year 2 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) Cohort 2
Number analyzed (Participants) | 264 | 259 | 264 | 57 | 57
Participants | 13 | 32 | 19 | 11 | 8
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs CHW - Cohort 2 vs Treatment as Usual (TAU) Cohort 2; Missing data at year 2 of intervention was imputed using MICE based on baseline characteristics and outcome values at year 1 of intervention. The statistical model was a mixed effects logistic regression with terms for the factorial design (TAU, AD, CHW, and cohort) and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Superiority; p = 0.032, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.71, 95% CI 2-sided [1.05 to 2.79]
Statistical Analysis 2: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs AD - Cohort 1 vs Treatment as Usual (TAU) Cohort 2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.376, Regression, Linear — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.68 to 2.75]
Statistical Analysis 3: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs Treatment as Usual (TAU) Cohort 2; Missing data at year 2 of intervention was imputed using MICE based on baseline characteristics and outcome values at year 1 of intervention. The statistical model was a mixed effects logistic regression with both additive terms and an interaction (TAU, AD, CHW, AD x CHW, and cohort) and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Other — Test of the additive assumption required by a factorial design. If the AD x CHW interaction is significant at p < 0.05, the additive assumption would have to be rejected; p = 0.645, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.42 to 4.05]

7. Secondary Outcome: Number of Participants Who Use of Any First Line, Evidence-based TUD Medication at the Intervention Year 1 or 2 Assessment in Cohorts 1 and 2
Description: Effects of CHW (pooled over AD+CHW and CHW) and AD (pooled over AD+CHW and AD) compared to usual care (TAU) on number of participants who use of any first line, evidence-based TUD medication during assessments for years 1 and 2 of the intervention. The investigators hypothesize that (1) those who receive CHW support will demonstrate higher rates of medication use than those who receive TAU, and (2) those with AD exposure will demonstrate higher rates of medication use than those who received TAU. To make use of all the data, hypotheses will be assessed in Cohorts 1 and 2 via analysis of a factorial design.
Time Frame: Any use over assessments for years 1 or 2 of intervention
Measure: Count of Participants; unit: Participants
Groups:
- Treatment as Usual (TAU) Cohort 2: Usual care (TAU) for adults with SMI in Massachusetts consists of rehabilitation services publicly funded by the state and traditional fee for service outpatient medical and psychiatric care. Importantly, medical care is not programmatically integrated with the psychiatric rehabilitation services. Participants in this arm will receive no other study-related intervention.Cohort 1 (AD-eligible) comprised participants seen in primary care clinics serving ≥3 enrolled participants. Cohort 2 (AD-ineligible) comprised participants whose primary care clinic served ≤2 enrolled participants
Arm/Group | Treatment as Usual (TAU) Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) Cohort 2
Number analyzed (Participants) | 264 | 259 | 264 | 57 | 57
Participants
  Any TUD medication | 112 | 121 | 83 | 30 | 24
  None | 152 | 138 | 181 | 27 | 33
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs CHW - Cohort 2 vs Treatment as Usual (TAU) Cohort 2; The statistical model was a mixed effects logistic regression with terms for the factorial design (TAU, AD, CHW, and cohort) and a clinic-varying random intercept; Test type: Superiority; p < 0.001, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; The CHW intervention increased odds of self-reported use of any TUD medication by 1.85; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.34 to 2.56]
Statistical Analysis 2: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs AD - Cohort 1 vs Treatment as Usual (TAU) Cohort 2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.084, Regression, Logistic; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.46 to 1.05]
Statistical Analysis 3: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs Treatment as Usual (TAU) Cohort 2; The statistical model was a mixed effects logistic regression with both additive terms and an interaction (TAU, AD, CHW, AD x CHW, and cohort) and a clinic-varying random intercept; Test type: Other — [test comment as in outcome 6, analysis 3]; p = 0.589, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.59 to 2.55]

8. Secondary Outcome: Number of Participants Who Use Varenicline at the Intervention Year 1 or 2 Assessments in Cohorts 1 and 2
Description: Effects of CHW (pooled over AD+CHW and CHW) and AD (pooled over AD+CHW and AD) compared to usual care (TAU) on number of participants who use varenicline during assessments for years 1 and 2 of the intervention. The investigators hypothesize that (1) those who receive CHW support will demonstrate higher rates of varenicline use than those who receive TAU, and (2) those with AD exposure will demonstrate higher rates of varenicline use than those who received TAU. To make use of all the data, hypotheses will be assessed in Cohorts 1 and 2 via analysis of a factorial design.
Time Frame: Any use over assessments for years 1 or 2 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) Cohort 2
Number analyzed (Participants) | 264 | 259 | 264 | 57 | 57
Participants
  Varenicline | 34 | 72 | 30 | 15 | 6
  Other | 230 | 187 | 234 | 42 | 51
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs CHW - Cohort 2 vs Treatment as Usual (TAU) Cohort 2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 3.05, 95% CI 2-sided [1.99 to 4.68]
Statistical Analysis 2: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs AD - Cohort 1 vs Treatment as Usual (TAU) Cohort 2; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.698, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.51 to 1.57]
Statistical Analysis 3: Comparison: Treatment as Usual (TAU) Cohort 1 vs AD + CHW - Cohort 1 vs Treatment as Usual (TAU) Cohort 2; [analysis description as in outcome 7, analysis 3]; Test type: Other — [test comment as in outcome 6, analysis 3]; p = 0.845, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.43 to 2.78]

9. Secondary Outcome: Effect of Use of Any TUD Medication on Number of Participants Who Are Abstinence at the Intervention Year 2 Assessment in Cohorts 1 and 2
Description: Effect of use of any first line, evidence-based TUD medication during assessments for years 1 and 2 of the intervention on number of participants who are abstinent (defined as 7-day point prevalence tobacco abstinence confirmed with an expired CO of 5 ppm or less) at the intervention year 2 assessment. The investigators hypothesize that those who used any medication will exhibit higher rates of tobacco abstinence than those who did not use any medications. To make use of all the data, the hypothesis will be assessed in Cohorts 1 and 2 via analysis of a factorial design. The indirect effect of CHW and AD interventions on abstinence rates with any TUD medication use as a mediator will be also be assessed.
Time Frame: Assessment at end of year 2 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) - Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) - Cohort 2
Number analyzed (Participants) | 264 | 259 | 264 | 57 | 57
Participants
  Any TUD med + abstinence | 5 | 24 | 7 | 7 | 2
  No TUD med + abstinence | 8 | 8 | 12 | 4 | 6
  Any TUD med + no abstinence | 107 | 100 | 78 | 23 | 22
  No TUD med + no abstinence | 144 | 127 | 167 | 23 | 27
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD + CHW - Cohort 1 vs AD - Cohort 1 vs CHW - Cohort 2 vs Treatment as Usual (TAU) - Cohort 2; Missing abstinence rates at year 2 of intervention were imputed using MICE based on baseline characteristics and abstinence rates at year 1 of intervention. The statistical model was a mixed effects logistic regression with terms for the factorial design (TAU, AD, CHW, and cohort) as well as TUD medication use and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Superiority; p = 0.158, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.92 to 2.20]; A mediation analysis found that the estimated proportion of the effect of TUD medication use on abstinence rates attributable to the CHW intervention was 55.6%

10. Secondary Outcome: Effect of Varenicline Use on Number of Participants Who Are Abstinence at the Intervention Year 2 Assessment in Cohorts 1 and 2
Description: Effect of use of varenicline during assessments for years 1 and 2 of the intervention on number of participants who are abstinent (defined as 7-day point prevalence tobacco abstinence confirmed with an expired CO of 5 ppm or less) at the intervention year 2 assessment. The investigators hypothesize that those who used varenicline will exhibit higher rates of tobacco abstinence than those who did not use any varenicline. To make use of all the data, the hypothesis will be assessed in Cohorts 1 and 2 via analysis of a factorial design. The indirect effect of CHW and AD interventions on abstinence rates with varenicline use as a mediator will be also be assessed.
Time Frame: Assessment at end of year 2 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) - Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) - Cohort 2
Number analyzed (Participants) | 264 | 259 | 264 | 57 | 57
Participants
  Varenicline + abstinence | 1 | 17 | 4 | 5 | 0
  No varenicline + abstinence | 12 | 15 | 15 | 6 | 8
  Varenicline + no abstinence | 33 | 55 | 26 | 10 | 6
  No varenicline + no abstinence | 218 | 172 | 219 | 36 | 43
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD + CHW - Cohort 1 vs AD - Cohort 1 vs CHW - Cohort 2 vs Treatment as Usual (TAU) - Cohort 2; Missing abstinence rates at year 2 of intervention were imputed using MICE based on baseline characteristics and abstinence rates at year 1 of intervention. The statistical model was a mixed effects logistic regression with terms for the factorial design (TAU, AD, CHW, and cohort) as well as varenicline use and a clinic-varying random intercept. Regression coefficients and mediation analysis estimates were pooled using Rubin's rule over 10 imputation runs; Test type: Superiority; p = 0.013, Regression, Logistic — The a priori threshold for significance was a p-value < 0.05; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.14 to 3.13]; A mediation analysis found that the estimated proportion of the effect of varenicline use on abstinence rates attributable to the CHW intervention was 36.6%

11. Secondary Outcome: Health-related Quality of Life Single-item Assessment at the Intervention Year 2 Assessment in Cohort 1
Description: Three pairwise comparisons between usual care (TAU), AD+CHW, and AD for health-related quality of life at the intervention year 2 assessment as assessed with the single-item self-reported Overall Health (SF-1) scale (measured on a 5-point scale from 1 = 'poor' to 5 = 'excellent'). The investigators hypothesize that (1) those who receive AD+CHW will demonstrate improved quality of life compared than those who receive TAU, (2) those who receive AD will demonstrate improved quality of life compared those who received TAU, and (3) those who receive AD+CHW will demonstrate improved quality of life compared than those who received AD.
Time Frame: Assessment at end of year 2 of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) - Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1
Number analyzed (Participants) | 252 | 248 | 253
score on a scale | 3.02 (0.96) | 3.13 (1.06) | 3.08 (0.99)
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD + CHW - Cohort 1; The model had a clinic varying random intercept. This statistical model included cohort 1: TAU , AD, and AD+CHW; Test type: Superiority; p = 0.505, Regression, Linear; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.16 to 0.33]
Statistical Analysis 2: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD - Cohort 1; Missing data at year 2 of intervention was imputed using MICE based on baseline characteristics and outcome values at year 1 of intervention. The statistical model was a mixed effects linear regression with terms for TAU, AD, and AD+CHW (cohort 1) and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Superiority; p = 0.848, Regression, Linear — The a priori threshold for significance was a p-value < 0.05; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.22 to 0.27]
Statistical Analysis 3: Comparison: AD + CHW - Cohort 1 vs AD - Cohort 1; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.529, Regression, Linear — The a priori threshold for significance was a p-value < 0.05; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.13 to 0.25]

12. Secondary Outcome: Health-related Quality of Life Single-item Assessment at the Intervention Year 2 Assessment in Cohorts 1 and 2
Description: Comparisons between (1) CHW (pooled over AD+CHW and CHW) and (2) AD (pooled over AD+CHW and AD) compared to usual care (TAU) on health-related quality of life at the intervention year 2 assessment as assessed with the single-item self-reported Overall Health (SF-1) scale (measured on a 5-point scale from 1 = 'poor' to 5 = 'excellent'). The investigators hypothesize that (1) those who receive CHW support will demonstrate improved quality of life compared to those who receive TAU, and (2) those with AD exposure will demonstrate improved quality of life compared to those who received TAU. To make use of all the data, hypotheses will be assessed in Cohorts 1 and 2 via analysis of a factorial design.
Time Frame: Assessment at end of year 2 of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) - Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) - Cohort 2
Number analyzed (Participants) | 252 | 248 | 253 | 53 | 55
score on a scale | 3.02 (0.96) | 3.13 (1.06) | 3.08 (0.99) | 3.11 (1.06) | 3.35 (0.90)
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD + CHW - Cohort 1 vs CHW - Cohort 2 vs Treatment as Usual (TAU) - Cohort 2; Missing data at year 2 of intervention was imputed using MICE based on baseline characteristics and outcome values at year 1 of intervention. The statistical model was a mixed effects linear regression with terms for the factorial design (TAU, AD, CHW, and cohort) and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Superiority; p = 0.937, Regression, Linear; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.16 to 0.18]
Statistical Analysis 2: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD + CHW - Cohort 1 vs AD - Cohort 1 vs Treatment as Usual (TAU) - Cohort 2; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.683, Regression, Linear; Median Difference (Final Values) = 0.05, 95% CI 2-sided [-0.19 to 0.29]
Statistical Analysis 3: Comparison: Treatment as Usual (TAU) - Cohort 1 vs AD + CHW - Cohort 1 vs Treatment as Usual (TAU) - Cohort 2; Missing data at year 2 of intervention was imputed using MICE based on baseline characteristics and outcome values at year 1 of intervention. The statistical model was a mixed effects linear regression with both additive terms and an interaction (TAU, AD, CHW, AD x CHW, and cohort) and a clinic-varying random intercept. Regression coefficients were pooled using Rubin's rule over 10 imputation runs; Test type: Other — [test comment as in outcome 6, analysis 3]; p = 0.190, Regression, Linear; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.15 to 0.74]

ADVERSE EVENTS:
Time Frame: 2 years
Description: We summarized the following adverse events comparing the intervention study arms: deceased, incarceration, med hospitalization, and psych hospitalization.
Groups:
- Treatment as Usual (TAU) - Cohort 2: Cohort 2 (AD-ineligible) comprised participants whose primary care clinic served ≤2 enrolled participants. Usual care (TAU) for adults with SMI in Massachusetts consists of rehabilitation services publicly funded by the state and traditional fee for service outpatient medical and psychiatric care. Importantly, medical care is not programmatically integrated with the psychiatric rehabilitation services. Participants in this arm will receive no other study-related intervention.
Arm/Group | Treatment as Usual (TAU) - Cohort 1 | AD + CHW - Cohort 1 | AD - Cohort 1 | CHW - Cohort 2 | Treatment as Usual (TAU) - Cohort 2
All-Cause Mortality (participants affected / at risk) | 14/333 | 18/336 | 16/341 | 3/78 | 0/77
Serious Adverse Events (participants affected / at risk) | 90/333 | 119/336 | 108/341 | 26/78 | 24/77
Other Adverse Events (participants affected / at risk) | 13/333 | 8/336 | 7/341 | 2/78 | 1/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (TAU) - Cohort 1 (N=333) | AD + CHW - Cohort 1 (N=336) | AD - Cohort 1 (N=341) | CHW - Cohort 2 (N=78) | Treatment as Usual (TAU) - Cohort 2 (N=77)
Medical hospitalization (General disorders) | 43 (77) | 59 (101) | 47 (97) | 10 (26) | 10 (22)
Psychiatric hospitalization (Psychiatric disorders) | 66 (168) | 82 (224) | 75 (182) | 19 (80) | 16 (45)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (TAU) - Cohort 1 (N=333) | AD + CHW - Cohort 1 (N=336) | AD - Cohort 1 (N=341) | CHW - Cohort 2 (N=78) | Treatment as Usual (TAU) - Cohort 2 (N=77)
Incarceration (Social circumstances) | 13 (13) | 8 (8) | 7 (7) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Annual survey didn't allow reliable discernment of sequenced monotherapies/combination therapy; Enrollment required SMI-related functional impairment severe enough for DMH-contracted psychiatric rehabilitation service eligibility; results may not generalize to individuals with SMI of lesser severity; Substantial loss to follow up, although no apparent differential dropout across randomization arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT02845440/Prot_SAP_001.pdf